CLINICAL TRIAL: NCT05737004
Title: The Effects of Prostate Cancer on Brain Function: a Prospective Cohort Study
Brief Title: Effects of Prostate Cancer on Brain Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EF2023-01
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; functional magnetic resonance imaging(fMRI); Brain function
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prostate cancer group: Prostate cancer was confirmed by biopsy, and fMRI examination 、Zung Self Rating Anxiety Scale and Beck Depression Inventory-II were performed in these patients within 1 week before biopsy .
  Interventions: Diagnostic Test: functional magnetic resonance imaging examination、Zung Self Rating Anxiety Scale and Beck Depression Inventory-II
- Non-Prostate cancer group: Non-Prostate cancer was confirmed by biopsy, and fMRI examination 、 Zung Self Rating Anxiety Scale and Beck Depression Inventory-II were performed in these patients within 1 week before biopsy .
  Interventions: Diagnostic Test: functional magnetic resonance imaging examination、Zung Self Rating Anxiety Scale and Beck Depression Inventory-II

INTERVENTIONS:
Diagnostic Test: functional magnetic resonance imaging examination、Zung Self Rating Anxiety Scale and Beck Depression Inventory-II — fMRI examination 、Zung Self Rating Anxiety Scale and Beck Depression Inventory-II were performed in these patients within 1 week before biopsy .

SUMMARY:
To explore whether the patients with prostate cancer have functional changes in specific brain areas and changes in psychological and mental characteristics compared with the patients without prostate cancer.

DETAILED DESCRIPTION:
This study was intended to observe the functional changes of brain fMRI in patients with and without prostate cancer enrolled in the cohort of patients who planned to undergo prostate biopsy, in an attempt to discover specific brain region changes in patients with prostate cancer, and lay a foundation for further clarifying the relationship and mechanism between brain region function changes and prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80
2. Patients with prostate biopsy;
3. No history of other malignant tumors;
4. Exclude other malignant tumors;
5. Fully understand the clinical trial protocol and sign informed consent;

Exclusion Criteria:

1. magnetic resonance contraindications;
2. symptomatic acute or chronic inflammation of the prostate;
3. Patients with brain trauma or brain disease;
4. Patients who have died of other malignancies in the past or are currently suffering from other malignancies;
5. Patients judged by the investigator to be unfit to participate in the clinical trial;

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient coming to our hospital for prostate biopsy and fully understand the clinical trial protocol and sign informed consent
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-04-13 (Estimated); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The evaluation of Magnetic Resonance(MR) | Within 1 week before biopsy
  To compare the differences in rs-fMRI measures (Amplitude of low frequency fluctuations , Regional Homogeneity and Functional Connectivity ) between prostate cancer group and Non-prostate cancer group.

SECONDARY OUTCOMES:
Assessment of anxiety status | Within 1 week before biopsy
  Zung Self Rating Anxiety Scale was used to assess anxiety status.By comparing the final score, less than or equal to 10 is considered healthy, and more than 10 is considered abnormal.
Assessment of depressive status | Within 1 week before biopsy
  Beck Depression Inventory-II was used to assess depressive status.By comparing the final scores, a score of 50 or less is considered healthy and a score of 50 or more is considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Once available, the results of this trial will be disseminated to an international peer-reviewed journal and presentations at international or national academic conferences. The data will be made available upon request to researchers a) who provide a methodologically sound proposal and b) whose proposed use of the data has been approved by an independent ethical review committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after publication with no end date